CLINICAL TRIAL: NCT01978899
Title: Healthy Living After Cancer: Weight Management Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Jennifer A. Ligibel, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-336
Record Dates: First submitted 2013-10-09; First posted 2013-11-08 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Weight Loss Program After Cancer Diagnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate Weight Loss Program Group (Active Comparator): Immediate Weight Loss Program Group
  * The weight loss Program Group will include weekly in-person sessions comprised of dietary counseling and increased physical activity. Patients will also be provided with exercise and dietary goals each week to implement at home.
  * Assessments will occur at baseline (pre-randomization), at the end of the 16-week intervention or control period and at 32 weeks.
  Interventions: Behavioral: Immediate Weight Loss Program Group
- Delayed Weight Loss Program Group (Active Comparator): The Delayed Weight Loss Program Group will take part in the weight loss intervention after the 16-week control period. Assessments will occur at baseline (pre-randomization), at the end of the 16-week intervention or control period and at 32 weeks
  Interventions: Behavioral: Delayed Weight Loss Program Group

INTERVENTIONS:
Behavioral: Immediate Weight Loss Program Group — Participation in 15-week Healthy Living Program.
  Arms: Immediate Weight Loss Program Group
Behavioral: Delayed Weight Loss Program Group — Participation in 15-week Healthy Living Program following 15-week wait period.
  Arms: Delayed Weight Loss Program Group

SUMMARY:
Studies have shown that patients who weigh more at the time of cancer diagnosis may be at increased risk of complications from surgery, fatigue, poor body image and other problems. Some research suggests that losing weight after cancer diagnosis can lead to improvements in these problems, as well as having other potential benefits for cancer survivors. Programs that reduce calories and increase exercise have been shown to help cancer survivors lose weight, but more research is needed to develop and test weight loss programs in cancer survivors.

This study is designed to look at the ability of a 15-week diet and exercise program to help cancer survivors lose weight. The investigator will look at changes in weight, body composition, quality of life, fatigue, body image as well as diet and exercise patterns, to see if this program can help men and women feel better and live healthier lives after cancer diagnosis.

DETAILED DESCRIPTION:
Before the research starts

* After signing this consent form, the participant will be asked to answer some questions about their health and ability to exercise to find out if the participant can be in the research study.
* If these tests show that the participant is eligible to participate in the research study, the participant will be able to participate in the research study. If the participant does not meet the eligibility criteria, the participant will not be able to participate in this research study.
* After the screening procedures confirm that the participant are eligible to participate in the research study.
* The participant will be scheduled to come to Dana-Farber to complete a number of study measures at baseline and at 16 and 32-weeks after the participant enrolls in the study.
* We will ask the participant to complete a number of study questionnaires that will include questions about: diet and exercise habits, medical history and quality of life (social support, thoughts and feelings).

It should take the participant about 30 minutes to complete the questionnaires. Some of the questions on these questionnaires are personal - the participant can refuse to answer these if the participant wishes. The information the participant provides is for research purposes only and will remain strictly confidential. The individuals (e.g. doctors, nurses, etc.) directly involved in the participant's care will not usually see their responses to these questions-if the participant wishes them to know this information please bring it to their attention.

Study staff will also record the participant's height and weight and will also ask the participant to undergo a walking test to measure how far the participant can comfortably walk in 6 minutes.

The participant will have an X-ray examination, called a dual energy x-ray absorptiometry (DEXA) scan that measures your body fat and bone mass at baseline and 16-weeks after enrollment. The DEXA scan involves lying still for about 10 minutes on a padded table. The scanner will not touch the participant and the participant will not feel any discomfort. The test does not require the participant to undress. If the participant wishes, we will provide your doctor with a copy of your DEXA scan.

Randomization (assignment to a group):

Because no one knows which of the study options is best, the participant will be "randomized" into one of the study groups: Immediate Weight Loss Program Group or Delayed Weight Loss Program Group. Randomization means that the participants are put into a group by chance. It is like flipping a coin. The central office that is coordinating the study will assign the participants to one of the two treatment groups. Neither the participant nor your doctor can choose what group the participant will be in. The participant will have an equal chance of being placed in either group.

Immediate Weight Loss Program Group If the participant is placed in the Immediate Weight Loss Program group, the participant will participate in the weight loss program soon after signing up for the study. The program consists of 15 sessions focused on reducing calories and increasing exercise. Sample goals of the program include reducing weight by 1-2 pounds per week and increasing exercise to at least 150 minutes of moderate exercise (such as walking) per week. Weight loss sessions will take place once per week for 15-weeks at Dana-Farber. The participant will meet with a dietician and exercise specialist weekly during the sessions to set diet and exercise goals for the week. Each session will consist of discussion of a diet and/or exercise topic for 30 minutes and 30 minutes of group exercise, such as moderate-paced walking or step aerobics. The participant will also be given the opportunity to be weighed, either as part of the group or in private with one of the weight loss study staff members, at each session in order to track their progress.

As part of participating in the weight loss program, the participant will be provided with a weight loss workbook with materials to supplement the weekly sessions. The participant will also be given a pedometer to help keep track of their exercise and a journal to keep track of their exercise and the food eaten each day. The participant will bring the journal to each weight loss session to review with study staff.

Delayed Weight Loss Program Group If the participant is placed in the Delayed Weight Loss Program group, he/or she will be offered the opportunity to participate in the weight loss program after an initial 15-week waiting period. During this waiting period, the participant is welcome to work on weight loss on your own, but the investigators will not provide the participant with the weight loss program materials or counseling until after the initial 15-week waiting period is over.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to any study-related procedures
* History of any malignancy
* Completed with all adjuvant surgery, chemotherapy and/or radiation at least one month prior to study enrollment (patients receiving ongoing hormonal or biologic therapy are eligible to participate)
* BMI >25kg/m2
* ECOG performance status of 0 or 1
* At least 18 years old
* Physically able to exercise and physician consent to start a weight loss program
* Willingness to be randomized
* English speaking and able to read English

Exclusion Criteria:

* Self-reported inability to walk 2 blocks (at any pace)
* Serious digestive and/or absorptive problems, including inflammatory bowel disease and chronic diarrhea that preclude adherence to the study diet.
* Bariatric surgery within the last year
* Cardiovascular, respiratory or musculoskeletal disease or joint problems that preclude moderate physical activity. Examples would include unstable angina, recent myocardial infarction, oxygen-dependent pulmonary disease, and osteoarthritis requiring imminent joint replacement. Moderate arthritis that does not preclude physical activity is not a reason for ineligibility.
* Psychiatric disorders or conditions that would preclude participation in the study intervention (e.g. untreated major depression or psychosis, substance abuse, severe personality disorder).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-11; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the impact of a 15-week, group-based weight loss intervention upon body weight in a group of cancer survivors. | 2 Years
  Change in weight (post-pre)weight loss intervention

SECONDARY OUTCOMES:
To evaluate the impact of a 15-week weight loss intervention upon the following in a group of cancer survivors. | 2 Years
  Correlate the effect of the intervention with anthropometric outcomes of percentage change or differences, changes in QOL, physical activity, or body image relative to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Ligibel, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to release individual participant data.

REFERENCES:
- [Derived] Brown JC, Giobbie-Hurder A, Yung RL, Mayer EL, Tolaney SM, Partridge AH, Ligibel JA. The effects of a clinic-based weight loss program on health-related quality of life and weight maintenance in cancer survivors: A randomized controlled trial. Psychooncology. 2022 Feb;31(2):326-333. doi: 10.1002/pon.5817. Epub 2021 Sep 12. PMID 34510643